CLINICAL TRIAL: NCT04707391
Title: A Phase IIIB, Randomized, Controlled, Observer-blind Study to Evaluate Safety and Immunogenicity of GSK's Meningococcal ABCWY Vaccine When Administered in Healthy Adolescents and Adults, Previously Primed With Meningococcal ACWY Vaccine
Brief Title: Immunogenicity and Safety Study of GSK's MenABCWY Vaccine in Healthy Adolescents and Adults Previously Primed With MenACWY Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 213171; 2019-004982-42 (EudraCT Number)
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Meningitis, Meningococcal
Keywords: Neisseria meningitidis; Meningococcal disease
MeSH Terms: conditions — Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines; 4CMenB vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ABCWY Group (Experimental): Participants received 2 doses of the MenABCWY vaccine on Day 1 and Day 181 (0,6-month schedule) and 1 dose of placebo on Day 211.
  Interventions: Combination Product: MenABCWY vaccine; Combination Product: Placebo
- ACWY Group (Active Comparator): Participants received 1 dose of MenACWY vaccine on Day 1 and 2 doses of MenB vaccine on Day 181 and Day 211.
  Interventions: Biological: MenACWY vaccine; Combination Product: MenB vaccine

INTERVENTIONS:
Combination Product: MenABCWY vaccine — 2 doses of MenABCWY vaccine administered intramuscularly on Day 1 and Day 181 to participants in ABCWY group.
  Arms: ABCWY Group
Combination Product: Placebo — 1 dose of placebo administered intramuscularly on Day 211 to participants in ABCWY group
  Arms: ABCWY Group
Biological: MenACWY vaccine — 1 dose of MenACWY vaccine administered intramuscularly on Day 1 to participants in ACWY group
  Other Names: Menveo
  Arms: ACWY Group
Combination Product: MenB vaccine — 2 doses of MenB vaccine administered intramuscularly on Day 181 and Day 211 to participants in ACWY group. MenB vaccine is a non-investigational medical product (NIMP) in this study and is administered only in compliance with standard of care.
  Other Names: Bexsero
  Arms: ACWY Group

SUMMARY:
The purpose of this study was to assess immunogenicity and safety of MenABCWY vaccine in healthy adolescents and adults aged 15 to 25 years previously vaccinated with MenACWY vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Participants and/or participants' parents/LARs, who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiary, return for follow-up visits).
2. Written or witnessed/thumb printed informed consent obtained from the participant/participant's parent(s)/LAR(s) of the participant prior to performance of any study specific procedure.
3. Written or witnessed/thumb printed informed assent obtained from participants below the legal age of consent prior to performance of any study specific procedure.
4. Previous vaccination with 1 dose of MenACWY vaccine at an age of 10 years or older, with an interval of at least 4 years between the previous MenACWY vaccine and enrollment (informed consent and assent [as applicable]) into this study.
5. A male or female between, and including, 15 and 25 years of age (i.e., 25 years and 364 days) at the time of the first vaccination.
6. Healthy participants as established by medical history, physical examination, and clinical judgment of the investigator before entering into the study.
7. Female participants of non-childbearing potential may be enrolled in the study. Non childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy, or post-menopause.
8. Female participants of childbearing potential may be enrolled in the study, if the participant:

   * has practiced adequate contraception for 30 days prior to vaccination, and
   * has a negative pregnancy test* on the day of vaccination, and
   * has agreed to continue adequate contraception during the entire intervention period and for 30 days after completion of the vaccination series.

Exclusion Criteria:

1. Current or previous, confirmed or suspected disease caused by N. meningitidis.
2. Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis infection within 60 days of enrollment.
3. History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s)/product.
4. Hypersensitivity, including allergy, to any component of vaccines, including diphtheria toxoid (CRM 197) and latex medicinal products or medical equipment whose use is foreseen in this study.
5. Progressive, unstable or uncontrolled clinical conditions
6. Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
7. Abnormal function or modification of the immune system resulting from:

   * Autoimmune disorders (including, but not limited to: blood, endocrine, hepatic, muscular, nervous system or skin autoimmune disorders; lupus erythematosus and associated conditions; rheumatoid arthritis and associated conditions; scleroderma and associated disorders) or immunodeficiency syndromes (including, but not limited to: acquired immunodeficiency syndromes and primary immunodeficiency syndromes).
   * Systemic administration of corticosteroids (oral/intravenous/intramuscular) for more than 14 consecutive days within 90 days prior to study vaccination until the following post vaccination blood sample. This will mean prednisone ≥20 mg/day (for adult participants and ≥0.5 mg/kg/day with maximum ≥20 mg/day for pediatric participants. Inhaled and topical steroids are allowed.
   * Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to study vaccination.
   * Administration of long-acting immune-modifying drugs at any time during the study period (e.g., infliximab).
8. Any neuroinflammatory (including but not limited to: demyelinating disorders, encephalitis or myelitis of any origin), congenital neurological conditions, encephalopathies, seizures (including all subtypes such as: absence seizures, generalized tonic-clonic seizures, partial complex seizures, partial simple seizures). History of febrile convulsions should not lead to exclusion.
9. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
10. Use of any investigational or non-registered product (drug, vaccine, or medical device) other than the study vaccine(s)/product during the period beginning 30 days before the first dose of study vaccine(s)/product (Day -29 to Day 1), or planned use during the study period.
11. Previous vaccination against any group B meningococcal vaccine at any time prior to informed consent and assent as applicable (according to the participant's age).
12. Previous vaccination with 2 or more doses of MenACWY vaccine.
13. Administration/planned administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before any dose of study vaccine(s)/product until the following post-vaccination blood sample.
14. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to any vaccine/product dose until the following post-vaccination blood sample. For corticosteroids, this will mean prednisone equivalent ≥20 mg/day for adult participants and ≥0.5 mg/kg/day with maximum ≥20 mg/day for pediatric participants. Inhaled and topical steroids are allowed.
15. Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non investigational vaccine/product (drug or medical device).
16. Child in care.
17. Pregnant or lactating female.
18. Female planning to become pregnant or planning to discontinue contraceptive precautions.
19. History of/current chronic alcohol and/or drug abuse.
20. Involvement in the study as a study staff member or being immediate dependents, family, or household member of a study staff member.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1250 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (45):
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Banning, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Sandy Springs, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Champaign, Illinois
  - GSK Investigational Site, Quincy, Illinois
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Methuen, Massachusetts
  - GSK Investigational Site, Roslindale, Massachusetts
  - GSK Investigational Site, Grosse Pointe Woods, Michigan
  - GSK Investigational Site, Biloxi, Mississippi
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Cranberry Township, Pennsylvania
  - GSK Investigational Site, Monongahela, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Carrollton, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Kaysville, Utah
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Seattle, Washington
- Argentina (7):
  - GSK Investigational Site, CABA, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Río Cuarto
- Australia (9):
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Kanwal, New South Wales
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Taringa, Queensland
  - GSK Investigational Site, Tarragindi, Queensland
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (3):
  - GSK Investigational Site, Guelph, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Nolan T, Bhusal C, Hoberman A, Llapur CJ, Voloshyna O, Fink E, Gentile A, Wallace G, Richmond PC, Domachowske JB, Mzolo T, Lattanzi M, Toneatto D; BOOST Study Group. Immunogenicity, Reactogenicity, and Safety of a Pentavalent Meningococcal ABCWY Vaccine in Adolescents and Young Adults Who Had Previously Received a Meningococcal ACWY Vaccine: A Phase 3, Randomized Controlled Clinical Study. Clin Infect Dis. 2025 Apr 30;80(4):752-760. doi: 10.1093/cid/ciae622. PMID 39722560

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 1250 participants enrolled,3 participants did not receive vaccination as they did not meet the eligibility criteria, therefore only 1247 participants were included in the Exposed Set and started the study.
Period: Overall Study
Arm/Group | ABCWY Group | ACWY Group
Started | 626 | 621
Completed | 541 | 542
Not Completed | 85 | 79
Not completed — Adverse Event | 5 | 8
Not completed — Lost to Follow-up | 44 | 31
Not completed — Protocol Violation | 1 | 5
Not completed — Withdrawal by Subject | 27 | 25
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 8 | 8
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABCWY Group | ACWY Group | Total
Number analyzed (Participants) | 626 | 621 | 1247
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 17.2 (2.53) | 17.2 (2.63) | 17.2 (2.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 343 | 324 | 667
  Male | 283 | 297 | 580
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 94 | 86 | 180
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 22 | 33 | 55
  Native Hawaiian or Other Pacific Islander | 2 | 6 | 8
  White | 474 | 464 | 938
  Other UNSPECIFIED | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Participants With a 4-fold Rise in Human Serum Bactericidal Assay (hSBA) Titers Against N. Meningitidis Serogroups A, C, W, and Y at 1 Month After the Second MenABCWY Vaccination and the Single MenACWY Vaccination, Relative to Baseline
Description: Four-fold rise is defined as: - a post-vaccination hSBA titer equal to or higher than (>=) 16 for participants with a pre-vaccination hSBA titer <4; - a post-vaccination hSBA titer >= 4 times the LLOQ for participants with a pre vaccination hSBA titer >= limit of detection (LOD) but < LLOQ; and - a post-vaccination hSBA titer >= 4 times the pre-vaccination titer for participants with a pre-vaccination hSBA titer >= LLOQ.
Time Frame: At 1 month after vaccination schedule (i.e., Day 211 for ABCWY group and Day 31 for ACWY group) compared to Day 1 (Baseline)
Population: Analysis was performed on Per Protocol Set (PPS), which included participants who received at least 1 dose of the study intervention to which they were randomized and had post-vaccination data available at the specified timepoint minus participants with protocol deviations that led to exclusion from the PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ABCWY Group | ACWY Group
Number analyzed (Participants) | 181 | 546
Percentage of Participants
  Meningitis A: number analyzed (Participants) | 169 | 505
  Meningitis A | 95.3 [90.89 to 97.93] | 95.0 [92.78 to 96.77]
  Meningitis C | 94.5 [90.07 to 97.32] | 94.0 [91.62 to 95.80]
  Meningitis W: number analyzed (Participants) | 181 | 544
  Meningitis W | 95.6 [91.48 to 98.07] | 93.9 [91.59 to 95.79]
  Meningitis Y: number analyzed (Participants) | 180 | 537
  Meningitis Y | 95.0 [90.72 to 97.69] | 94.4 [92.12 to 96.20]
Statistical Analysis 1: Comparison: ABCWY Group vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with a MenACWY vaccine, as measured by the percentages of participants achieving a 4-fold rise in hSBA titers against N. meningitidis serogroups A at 1 month after the second MenABCWY vaccination (0,6-months) and 1 month after the MenACWY vaccination (single dose); Test type: Non-Inferiority — Non-inferiority was to be demonstrated if the lower limit of the two-sided 95% Confidence Interval(CI) for the difference in percenatge of participants achieving a 4-fold rise in hSBA titers between MenABCWY group and MenACWY group was above -10% for serogroup A; Difference in percentage of participants = 0.2, 0.95% CI 2-sided [-4.38 to 3.50]
Statistical Analysis 2: Comparison: ABCWY Group vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with a MenACWY vaccine, as measured by the percentages of participants achieving a 4-fold rise in hSBA titers against N. meningitidis serogroups C at 1 month after the second MenABCWY vaccination (0,6-months) and 1 month after the MenACWY vaccination (single dose); Test type: Non-Inferiority — Non-inferiority was to be demonstrated if the lower limit of the two-sided 95% Confidence Interval(CI) for the difference in percenatge of participants achieving a 4-fold rise in hSBA titers between MenABCWY group and MenACWY group was above -10% for serogroup C; Difference in percentage of participants = 0.5, 0.95% CI 2-sided [-4.14 to 3.98]
Statistical Analysis 3: Comparison: ABCWY Group vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with a MenACWY vaccine, as measured by the percentages of participants achieving a 4-fold rise in hSBA titers against N. meningitidis serogroups W at 1 month after the second MenABCWY vaccination (0,6-months) and 1 month after the MenACWY vaccination (single dose); Test type: Non-Inferiority — Non-inferiority was to be demonstrated if the lower limit of the two-sided 95% Confidence Interval(CI) for the difference in percenatge of participants achieving a 4-fold rise in hSBA titers between MenABCWY group and MenACWY group was above -10% for each serogroup W; Difference in percentage of participants = 1.6, 0.95% CI 2-sided [-2.73 to 4.89]
Statistical Analysis 4: Comparison: ABCWY Group vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with a MenACWY vaccine, as measured by the percentages of participants achieving a 4-fold rise in hSBA titers against N. meningitidis serogroups Y at 1 month after the second MenABCWY vaccination (0,6-months) and 1 month after the MenACWY vaccination (single dose); Test type: Non-Inferiority — Non-inferiority was to be demonstrated if the lower limit of the two-sided 95% Confidence Interval(CI) for the difference in percenatge of participants achieving a 4-fold rise in hSBA titers between MenABCWY group and MenACWY group was above -10% for each serogroup Y; Difference in percentage of participants = 0.6, 0.95% CI 2-sided [-3.93 to 3.91]

2. Primary Outcome: Percentages of Participants With a 4-fold Rise in hSBA Titers Against N. Meningitidis Serogroups A, C, W, and Y at 1 Month After the First MenABCWY Vaccination and the Single MenACWY Vaccination, Relative to Baseline
Description: as for outcome 1
Time Frame: At 1 month after the first vaccination (i.e., Day 31) compared to Day 1 (Baseline)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ABCWY Group | ACWY Group
Number analyzed (Participants) | 570 | 546
Percentage of Participants
  Meningitis A: number analyzed (Participants) | 509 | 505
  Meningitis A | 92.5 [89.90 to 94.66] | 95.0 [92.78 to 96.77]
  Meningitis C | 94.0 [91.76 to 95.83] | 94.0 [91.62 to 95.80]
  Meningitis W: number analyzed (Participants) | 565 | 544
  Meningitis W | 94.3 [92.10 to 96.09] | 93.9 [91.59 to 95.79]
  Meningitis Y: number analyzed (Participants) | 567 | 537
  Meningitis Y | 93.7 [91.32 to 95.51] | 94.4 [92.12 to 96.20]
Statistical Analysis 1: Comparison: ABCWY Group vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with a MenACWY vaccine, as measured by the percentages of participants achieving a 4-fold rise in hSBA titers against N. meningitidis serogroups A at 1 month after the first MenABCWY vaccination (0,6-months) and 1 month after the MenACWY vaccination (single dose); Test type: Non-Inferiority — Non-inferiority was to be demonstrated if the lower limit of the two-sided 95% Confidence Interval(CI) for the difference in percenatge of participants achieving a 4-fold rise in the 4-fold rise in hSBA titers (p_MenABCWY- p_MenACWY) is above -10% for serogroup A; Difference in percentage of participants = -2.5, 0.95% CI 2-sided [-5.59 to 0.47]
Statistical Analysis 2: Comparison: ABCWY Group vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with a MenACWY vaccine, as measured by the percentages of participants achieving a 4-fold rise in hSBA titers against N. meningitidis serogroups C at 1 month after the first MenABCWY vaccination (0,6-months) and 1 month after the MenACWY vaccination (single dose); Test type: Non-Inferiority — Non-inferiority was to be demonstrated if the lower limit of the two-sided 95% Confidence Interval(CI) for the difference in percenatge of participants achieving a 4-fold rise in hSBA titers (p_MenABCWY- p_MenACWY) is above -10% for serogroup C; Difference in percentage of participants = 0.1, 0.95% CI 2-sided [-2.76 to 2.94]
Statistical Analysis 3: Comparison: ABCWY Group vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with a MenACWY vaccine, as measured by the percentages of participants achieving a 4-fold rise in hSBA titers against N. meningitidis serogroupsW at 1 month after the first MenABCWY vaccination (0,6-months) and 1 month after the MenACWY vaccination (single dose); Test type: Non-Inferiority — Non-inferiority was to be demonstrated if the lower limit of the two-sided 95% Confidence Interval(CI) for the difference in percenatge of participants achieving a 4-fold rise in hSBA titers (p_MenABCWY- p_MenACWY) is above -10% for serogroup W; Difference in percentage of participants = 0.4, 0.95% CI 2-sided [-2.41 to 3.25]
Statistical Analysis 4: Comparison: ABCWY Group vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with a MenACWY vaccine, as measured by the percentages of participants achieving a 4-fold rise in hSBA titers against N. meningitidis serogroups Y at 1 month after the first MenABCWY vaccination (0,6-months) and 1 month after the MenACWY vaccination (single dose); Test type: Non-Inferiority — Non-inferiority was to be demonstrated if the lower limit of the two-sided 95% Confidence Interval(CI) for the difference in percenatge of participants achieving a 4-fold rise in hSBA titers (p_MenABCWY- p_MenACWY) is above -10% for serogroup Y; Difference in percentage of participants = -0.8, 0.95% CI 2-sided [-3.62 to 2.09]

3. Primary Outcome: Number of Participants With Solicited Administration Site Events Following Vaccination at Day 1 for ABCWY Group and ACWY Group
Description: Assessed solicited administration site events include injection site pain, erythema, swelling, induration. Any pain = occurrence of the symptom regardless of intensity grade and any erythema, swelling and induration are defined as a symptom with a surface diameter equal to or greater than 25 millimeters.
Time Frame: During the 7 days (including day of vaccination) following vaccination at day 1 for ABCWY group and ACWY group
Population: Analysis was performed on Solicited Safety Set (SSS),which included participants who received at least 1 dose of the study intervention and had solicited administration data available during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Group | ACWY Group
Number analyzed (Participants) | 608 | 601
Participants
  Injection site pain | 486 | 191
  Erythema: number analyzed (Participants) | 608 | 600
  Erythema | 29 | 9
  Swelling: number analyzed (Participants) | 608 | 600
  Swelling | 26 | 13
  Induration: number analyzed (Participants) | 608 | 600
  Induration | 24 | 14

4. Primary Outcome: Number of Participants With Solicited Administration Site Events Following Vaccination at Day 181 for ABCWY Group
Description: as for outcome 3
Time Frame: During the 7 days (including day of vaccination) following vaccination at Day 181 for ABCWY group
Population: Analysis was performed on Solicited Safety Set (SSS), which included participants who received at least 2 dose of the study intervention and had solicited data available during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Group
Number analyzed (Participants) | 507
Participants
  Injection site pain | 377
  Erythema: number analyzed (Participants) | 505
  Erythema | 31
  Swelling: number analyzed (Participants) | 505
  Swelling | 30
  Induration: number analyzed (Participants) | 505
  Induration | 22

5. Primary Outcome: Number of Participants With Solicited Systemic Events Following Vaccination at Day 1 for the ABCWY Group and ACWY Group
Description: Assessed solicited systemic events include fever [body temperature >= 38.0°C (celsius) /100.4°F (Fahrenheit)], nausea, fatigue, myalgia, arthralgia, headache.
Time Frame: During the 7 days (including day of vaccination) following vaccination at day 1 for the ABCWY group and ACWY group
Population: Analysis was performed on Solicited Safety Set (SSS), which included participants who received at least 1 dose of the study intervention and had solicited systemic data available during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Group | ACWY Group
Number analyzed (Participants) | 608 | 601
Participants
  Fever: number analyzed (Participants) | 608 | 600
  Fever | 12 | 7
  Nausea: number analyzed (Participants) | 608 | 600
  Nausea | 88 | 75
  Fatigue: number analyzed (Participants) | 608 | 600
  Fatigue | 244 | 222
  Myalgia: number analyzed (Participants) | 608 | 600
  Myalgia | 90 | 66
  Arthralgia: number analyzed (Participants) | 608 | 600
  Arthralgia | 45 | 49
  Headache | 249 | 208

6. Primary Outcome: Number of Participants With Solicited Systemic Events Following Vaccination at Day 181 for the ABCWY Group
Description: Assessed solicited systemic events include fever [body temperature >= 38.0°C/100.4°F], nausea, fatigue, myalgia, arthralgia, headache.
Time Frame: During the 7 days (including day of vaccination) following vaccination at day 181 for the ABCWY group
Population: Analysis was performed on Solicited Safety Set (SSS),which included participants who received at least 2 dose of the study intervention and had solicited systemic data available during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Group
Number analyzed (Participants) | 505
Participants
  Fever | 9
  Nausea | 58
  Fatigue | 167
  Myalgia | 67
  Arthralgia | 30
  Headache | 167

7. Primary Outcome: Number of Participants With Any Unsolicited Adverse Events (AEs) (Including All Serious Adverse Events [SAEs], AEs Leading to Withdrawal, AEs of Special Interest [AESIs] and Medically Attended AEs)
Description: Unsolicited AE-AE not solicited using an eDiary and spontaneously communicated by a participant/participant's parent(s)/Legally acceptable representative(s) who has signed informed consent. SAEs-events that result in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is congenital anomaly/birth defect in the offspring of a study participant/results in abnormal pregnancy outcomes. AESIs-predefined AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation in order to characterize and understand it. An MAE is defined as an unsolicited AE for which the participant received medical attention such as hospitalization, or an emergency room visit, or visit to/by a health care provider.
Time Frame: During the 30 days (including day of vaccination) following vaccination at day 1 for ABCWY group and ACWY group
Population: Analysis was performed on the Unsolicited Safety Set (USS), which included participants who received at least 1 dose of the study intervention and had unsolicited AEs during the specific period.
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Group | ACWY Group
Number analyzed (Participants) | 626 | 621
Participants | 96 | 93

8. Primary Outcome: Number of Participants With Any Unsolicited Adverse Events (AEs) (Including All Serious Adverse Events [SAEs], AEs Leading to Withdrawal, AEs of Special Interest [AESIs] and Medically Attended AEs) Following Vaccination at Day 181 for ABCWY Group
Description: Any AE-untoward medical occurrence in a patient/clinical investigation participant, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. Unsolicited AE-AE not solicited using an eDiary and spontaneously communicated by a participant/participant's parent(s)/Legally acceptable representative(s) who has signed informed consent. SAEs-events that result in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is congenital anomaly/birth defect in the offspring of a study participant/results in abnormal pregnancy outcomes. AESIs-predefined AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation in order to characterize and understand it.
Time Frame: During the 30 days (including day of vaccination) following vaccination at day 181 for ABCWY group
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Group
Number analyzed (Participants) | 626
Participants | 72

9. Primary Outcome: Number of Participants With SAEs, AEs Leading to Withdrawal, AESIs and Medically Attended AEs
Description: SAEs, AEs leading to withdrawal, AESIs and medically attended AEs were assessed throughout the study period are reported in this outcome measure.
Time Frame: From Day 1 to Day 361 (throughout the study period)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY Group | ACWY Group
Number analyzed (Participants) | 626 | 621
Participants
  SAEs | 18 | 7
  AEs leading to withdrawal | 4 | 6
  AESIs | 0 | 4
  Medically Attended AEs | 223 | 206

10. Secondary Outcome: Percentages of Participants With hSBA Titers >= Lower Limit of Quantitation (LLOQ) Against Serogroups A, C, W, and Y at Day 1, 1 Month After the First MenABCWY Vaccination and After the Single MenACWY Vaccination
Description: The immune response to MenABCWY vaccine after the first dose and single dose of MenACWY vaccine was evaluated by measuring the percentage of participants with hSBA titers >= LLOQ against each of the serogroups A, C, W and Y.
Time Frame: At Day 1 (pre-vaccination) and 1 month after the vaccination schedule (i.e., Day 31 for ABCWY group [first dose] and ACWY group)
Population: Analysis was performed on the Full Analysis Set (FAS), which included participants who received at least 1 dose of the study intervention and had post-vaccination immunogenicity data for the specified analysis at the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ABCWY Group | ACWY Group
Number analyzed (Participants) | 609 | 593
Percentage of Participants
  Meningitis A, Day 1: number analyzed (Participants) | 546 | 549
  Meningitis A, Day 1 | 27.7 [23.94 to 31.61] | 28.8 [25.02 to 32.77]
  Meningitis A, Day 31: number analyzed (Participants) | 605 | 585
  Meningitis A, Day 31 | 98.3 [96.98 to 99.20] | 98.1 [96.66 to 99.06]
  Meningitis C, Day 1: number analyzed (Participants) | 601 | 584
  Meningitis C, Day 1 | 57.7 [53.67 to 61.72] | 56.2 [52.03 to 60.23]
  Meningitis C, Day 31 | 98.9 [97.65 to 99.54] | 99.0 [97.81 to 99.63]
  Meningitis W, Day 1: number analyzed (Participants) | 597 | 583
  Meningitis W, Day 1 | 36.3 [32.48 to 40.35] | 33.4 [29.62 to 37.44]
  Meningitis W, Day 31: number analyzed (Participants) | 607 | 592
  Meningitis W, Day 31 | 98.4 [96.99 to 99.21] | 96.8 [95.03 to 98.06]
  Meningitis Y, Day 1: number analyzed (Participants) | 600 | 576
  Meningitis Y, Day 1 | 37.5 [33.61 to 41.51] | 34.9 [31.00 to 38.94]
  Meningitis Y, Day 31: number analyzed (Participants) | 606 | 591
  Meningitis Y, Day 31 | 97.9 [96.36 to 98.85] | 97.6 [96.06 to 98.70]

11. Secondary Outcome: Percentages of Participants With hSBA Titers >= Lower Limit of Quantitation (LLOQ) Against Serogroups A, C, W, and Y at 1 Month After the Second MenABCWY Vaccination
Description: The immune response to MenABCWY vaccine after the second dose was evaluated by measuring the percentage of participants with hSBA titers >= LLOQ against each of the serogroups A, C, W and Y.
Time Frame: 1 month after the vaccination schedule (i.e., Day 211 for ABCWY group [second dose])
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ABCWY Group
Number analyzed (Participants) | 609
Percentage of Participants
  Meningitis A, Day 211: number analyzed (Participants) | 213
  Meningitis A, Day 211 | 99.5 [97.41 to 99.99]
  Meningitis C, Day 211: number analyzed (Participants) | 211
  Meningitis C, Day 211 | 100.0 [98.27 to 100.00]
  Meningitis W, Day 211: number analyzed (Participants) | 212
  Meningitis W, Day 211 | 100.0 [98.28 to 100.00]
  Meningitis Y, Day 211: number analyzed (Participants) | 210
  Meningitis Y, Day 211 | 100.0 [98.26 to 100.00]

12. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Against Serogroups A, C, W, and Y at Day 1, 1 Month After the First MenABCWY Vaccination and After the Single MenACWY Vaccination
Description: The immune response to MenABCWY after first dose and single dose of MenACWY vaccine was evaluated by measuring the human serum bactericidal activity against each of the serogroups A, C, W and Y in terms of GMTs. For each serogroup, the GMTs with their associated 2-sided 95% confidence intervals were calculated.
Time Frame: At Day 1 and 1 month after the vaccination schedule (i.e., Day 31 for ABCWY group [first dose] and ACWY group)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY Group | ACWY Group
Number analyzed (Participants) | 609 | 593
Titers
  Meningitis A, Day 1: number analyzed (Participants) | 546 | 549
  Meningitis A, Day 1 | 15.30 [13.07 to 17.92] | 16.34 [13.96 to 19.14]
  Meningitis A, Day 31: number analyzed (Participants) | 605 | 585
  Meningitis A, Day 31 | 670.78 [594.71 to 756.58] | 1282.56 [1135.84 to 1448.23]
  Meningitis C, Day 1: number analyzed (Participants) | 601 | 584
  Meningitis C, Day 1 | 31.90 [26.63 to 38.23] | 29.76 [24.81 to 35.71]
  Meningitis C, Day 31 | 2945.68 [2471.13 to 3511.36] | 2552.27 [2138.66 to 3045.87]
  Meningitis W, Day 1: number analyzed (Participants) | 597 | 583
  Meningitis W, Day 1 | 12.08 [10.31 to 14.15] | 11.08 [9.45 to 12.99]
  Meningitis W, Day 31: number analyzed (Participants) | 607 | 592
  Meningitis W, Day 31 | 1899.60 [1638.73 to 2202.00] | 1665.64 [1435.57 to 1932.58]
  Meningitis Y, Day 1: number analyzed (Participants) | 600 | 576
  Meningitis Y, Day 1 | 12.84 [11.16 to 14.76] | 11.86 [10.29 to 13.66]
  Meningitis Y, Day 31: number analyzed (Participants) | 606 | 591
  Meningitis Y, Day 31 | 1590.71 [1380.78 to 1832.55] | 1578.42 [1369.00 to 1819.88]

13. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Against Serogroups A, C, W, and Y at 1 Month After the Second MenABCWY Vaccination
Description: The immune response to MenABCWY after second dose was evaluated by measuring the human serum bactericidal activity against each of the serogroups A, C, W and Y in terms of GMTs. For each serogroup, the GMTs with their associated 2-sided 95% confidence intervals were calculated.
Time Frame: 1 month after the vaccination schedule (i.e., Day 211 for ABCWY group [second dose])
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY Group
Number analyzed (Participants) | 609
Titers
  Meningitis A, Day 211: number analyzed (Participants) | 213
  Meningitis A, Day 211 | 645.24 [544.11 to 765.16]
  Meningitis C, Day 211: number analyzed (Participants) | 211
  Meningitis C, Day 211 | 2350.14 [1809.69 to 3052.00]
  Meningitis W, Day 211: number analyzed (Participants) | 212
  Meningitis W, Day 211 | 1173.61 [940.25 to 1464.89]
  Meningitis Y, Day 211: number analyzed (Participants) | 210
  Meningitis Y, Day 211 | 1130.54 [916.85 to 1394.04]

14. Secondary Outcome: Geometric Mean Ratios (GMRs) Against Serogroups A, C, W, and Y at 1 Month After the First MenABCWY Vaccination and After the Single MenACWY Vaccination
Description: The immune response to MenABCWY vaccine after first and single dose of MenACWY vaccine are evaluated by measuring the human serum bactericidal activity against each of the serogroups A, C, W and Y, compared to baseline (Day 1) and expressed as GMRs. Within group GMRs was calculated as ratio of GMTs in the post-vaccination timepoint to the pre-vaccination timepoint.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 31 for ABCWY group [first dose] and ACWY group) compared to baseline (Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ABCWY Group | ACWY Group
Number analyzed (Participants) | 597 | 583
Ratio
  Meningitis A, Day 31: number analyzed (Participants) | 539 | 539
  Meningitis A, Day 31 | 43.98 [36.92 to 52.40] | 76.91 [64.53 to 91.66]
  Meningitis C, Day 31 | 92.87 [77.13 to 111.83] | 86.36 [71.63 to 104.12]
  Meningitis W, Day 31: number analyzed (Participants) | 591 | 581
  Meningitis W, Day 31 | 154.09 [125.80 to 188.73] | 150.83 [123.00 to 184.96]
  Meningitis Y, Day 31: number analyzed (Participants) | 593 | 573
  Meningitis Y, Day 31 | 124.11 [103.23 to 149.23] | 134.66 [111.75 to 162.26]

15. Secondary Outcome: Geometric Mean Ratios (GMRs) Against Serogroups A, C, W, and Y at 1 Month After Second MenABCWY Vaccination
Description: The immune response to MenABCWY vaccine after second dose are evaluated by measuring the human serum bactericidal activity against each of the serogroups A, C, W and Y, compared to baseline (Day 1) and expressed as GMRs. Within group GMRs was calculated as ratio of GMTs in the post-vaccination timepoint to the pre-vaccination timepoint.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 211 for ABCWY group [second dose]) compared to baseline (Day 1)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ABCWY Group
Number analyzed (Participants) | 597
Ratio
  Meningitis A, Day 211: number analyzed (Participants) | 196
  Meningitis A, Day 211 | 44.74 [34.67 to 57.74]
  Meningitis C, Day 211: number analyzed (Participants) | 205
  Meningitis C, Day 211 | 68.33 [52.19 to 89.46]
  Meningitis W, Day 211: number analyzed (Participants) | 207
  Meningitis W, Day 211 | 97.66 [72.52 to 131.52]
  Meningitis Y, Day 211: number analyzed (Participants) | 202
  Meningitis Y, Day 211 | 82.45 [62.80 to 108.24]

16. Secondary Outcome: Percentages of Participants With hSBA Titers >= LLOQ for Each and All Serogroup B Indicator Strains at Day 1 and at 1 Month After the Second Dose of MenABCWY Vaccination
Description: The immune response to MenABCWY vaccine after second dose was evaluated by measuring bactericidal activity against each (individual response) and all (composite response) N. meningitidis serogroup B indicator strains (M14459, 96217, M13520 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively).
Time Frame: At Day 1 and at Day 211
Population: Analysis was performed on the Full Analysis Set (FAS), which included participants from only ABCWY Group who received at least 1 dose of the MenABCWY vaccine and had post vaccination immunogenicity data for the specified analysis at the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ABCWY Group
Number analyzed (Participants) | 184
Percentage of Participants
  fHbp (M14459) Ab, Day 1 | 8.7 [5.05 to 13.74]
  fHbp (M14459) Ab, Day 211: number analyzed (Participants) | 165
  fHbp (M14459) Ab, Day 211 | 88.5 [82.60 to 92.92]
  NadA (96217) Ab, Day 1: number analyzed (Participants) | 183
  NadA (96217) Ab, Day 1 | 7.7 [4.25 to 12.50]
  NadA (96217) Ab, Day 211: number analyzed (Participants) | 165
  NadA (96217) Ab, Day 211 | 95.8 [91.45 to 98.28]
  NHBA (M13520) Ab, Day 1: number analyzed (Participants) | 183
  NHBA (M13520) Ab, Day 1 | 20.2 [14.65 to 26.77]
  NHBA (M13520) Ab, Day 211: number analyzed (Participants) | 164
  NHBA (M13520) Ab, Day 211 | 96.3 [92.21 to 98.65]
  PorAP1.4 (NZ98/254) Ab, Day 1 | 2.7 [0.89 to 6.23]
  PorAP1.4 (NZ98/254) Ab, Day 211: number analyzed (Participants) | 164
  PorAP1.4 (NZ98/254) Ab, Day 211 | 75.6 [68.30 to 81.97]
  Composite Response, Day 1: number analyzed (Participants) | 181
  Composite Response, Day 1 | 1.1 [0.13 to 3.93]
  Composite Response, Day 211: number analyzed (Participants) | 164
  Composite Response, Day 211 | 72.0 [64.41 to 78.68]

17. Secondary Outcome: Percentages of Participants With 4-fold Rise in hSBA Titers Against Each N. Meningitidis Serogroup B Indicator Strains at 1 Month After the Second MenABCWY Vaccination
Description: The immune response to MenABCWY after second dose is evaluated by measuring bactericidal activity against each of the N. meningitidis serogroup B test strains (M14459, 96217, M13520 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively). compared to baseline (day 1) in terms of 4-fold rise in hSBA titers. For each of the serogroup B indicator strains, the 4-fold rise is defined as: a post-vaccination hSBA titer >=16 for participants with a pre-vaccination hSBA titer <4; . a post-vaccination hSBA titer >= 4 times the LLOQ for participants with a prevaccination hSBA titer >= limit of detection (LOD) but < LLOQ; and, a post-vaccination hSBA titer >= 4 times the pre-vaccination titer for participants with a pre-vaccination hSBA titer >= LLOQ.
Time Frame: At Day 211 compared to baseline (Day 1)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ABCWY Group
Number analyzed (Participants) | 163
Percentage of Participants
  fHbp (M14459) Ab | 68.1 [60.35 to 75.17]
  NadA (96217) Ab: number analyzed (Participants) | 162
  NadA (96217) Ab | 90.1 [84.46 to 94.25]
  NHBA (M13520) Ab: number analyzed (Participants) | 161
  NHBA (M13520) Ab | 64.6 [56.68 to 71.96]
  PorAP1.4 (NZ98/254) Ab: number analyzed (Participants) | 162
  PorAP1.4 (NZ98/254) Ab | 45.7 [37.84 to 53.68]

18. Secondary Outcome: GMTs Against Each Serogroup B Indicator Strains at Day 1 and at 1 Month After Second MenABCWY Vaccination
Description: The immune response to MenABCWY vaccine after the second dose was evaluated by measuring bactericidal activity against each of the N. meningitidis serogroup B indicator strains (M14459, 96217, M13520 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively) in terms of GMTs at baseline (Day 1) and 1 month after second MenABCWY vaccination.
Time Frame: At Day 1 and at Day 211
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY Group
Number analyzed (Participants) | 184
Titers
  fHbp (M14459) Ab, Day 1 | 2.84 [2.53 to 3.19]
  fHbp (M14459) Ab, Day 211: number analyzed (Participants) | 165
  fHbp (M14459) Ab, Day 211 | 17.56 [13.52 to 22.80]
  NadA (96217) Ab, Day 1: number analyzed (Participants) | 183
  NadA (96217) Ab, Day 1 | 8.62 [7.39 to 10.06]
  NadA (96217) Ab, Day 211: number analyzed (Participants) | 165
  NadA (96217) Ab, Day 211 | 143.61 [106.71 to 193.26]
  NHBA (M13520) Ab, Day 1: number analyzed (Participants) | 183
  NHBA (M13520) Ab, Day 1 | 3.28 [2.59 to 4.15]
  NHBA (M13520) Ab, Day 211: number analyzed (Participants) | 164
  NHBA (M13520) Ab, Day 211 | 24.82 [19.19 to 32.11]
  PorAP1.4 (NZ98/254) Ab, Day 1 | 3.13 [2.86 to 3.43]
  PorAP1.4 (NZ98/254) Ab, Day 211: number analyzed (Participants) | 164
  PorAP1.4 (NZ98/254) Ab, Day 211 | 11.44 [8.61 to 15.19]

19. Secondary Outcome: GMRs Against Each Serogroup B Indicator Strains at 1 Month After Second Dose of MenABCWY Vaccination
Description: The immune response to MenABCWY vaccine after second dose was evaluated by measuring the human serum bactericidal activity against each of the N. meningitidis serogroup B indicator strains (M14459, 96217, M13520 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively) compared to baseline (Day 1) and expressed as GMRs. Within group GMRs was calculated as ratio of GMTs in the post-vaccination timepoint to the pre-vaccination timepoint.
Time Frame: At Day 211 compared to baseline (Day 1)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ABCWY Group
Number analyzed (Participants) | 163
Ratio
  fHbp (M14459) Ab | 6.29 [4.84 to 8.18]
  NadA (96217) Ab: number analyzed (Participants) | 162
  NadA (96217) Ab | 16.67 [12.25 to 22.70]
  NHBA (M13520) Ab: number analyzed (Participants) | 161
  NHBA (M13520) Ab | 7.69 [6.08 to 9.72]
  PorAP1.4 (NZ98/254) Ab: number analyzed (Participants) | 162
  PorAP1.4 (NZ98/254) Ab | 3.65 [2.76 to 4.83]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during the 7-day follow-up period after vaccination. Unsolicited AEs were collected during the 30-day follow-up period after vaccination. SAEs were collected through the entire period of the study (from Day 1 up to study end [Day 361])
Arm/Group | ABCWY Group | ACWY Group
All-Cause Mortality (participants affected / at risk) | 1/626 | 1/621
Serious Adverse Events (participants affected / at risk) | 18/626 | 7/621
Other Adverse Events (participants affected / at risk) | 583/626 | 552/621
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABCWY Group (N=626) | ACWY Group (N=621)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal disease (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Gastroschisis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Wolff-Parkinson-White syndrome congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABCWY Group (N=626) | ACWY Group (N=621)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 3 (3) | 6 (6)
Atypical pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (3)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cervicitis human papilloma virus (Infections and infestations) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 5 (5) | 2 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 92 (97) | 97 (99)
Cystitis (Infections and infestations) | 2 (3) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 2 (2)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal foot infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Gonorrhoea (Infections and infestations) | 2 (3) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Herpeszoster (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 3 (3) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 11 (11) | 7 (7)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis viral (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 10 (11) | 6 (6)
Omphalitis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 2 (2) | 3 (3)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 2 (2) | 3 (3)
Paronychia (Infections and infestations) | 2 (2) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Pericoronitis (Infections and infestations) | 0 (0) | 2 (3)
Pharyngitis (Infections and infestations) | 5 (5) | 7 (8)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 7 (7) | 6 (6)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal disease (Infections and infestations) | 2 (3) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 2 (2)
Pyuria (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5) | 10 (10)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2)
Trichomoniasis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 17 (17) | 8 (8)
Urinary tract infection (Infections and infestations) | 10 (10) | 7 (7)
Viral infection (Infections and infestations) | 1 (1) | 4 (4)
Viral pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 7 (8) | 9 (9)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Infected naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypocomplementaemia (Immune system disorders) | 0 (0) | 1 (1)
Mite allergy (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 6 (6) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 13 (13) | 8 (8)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 5 (5) | 4 (4)
Autism spectrum disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Behavioural insomnia of childhood (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Borderline personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 7 (8) | 8 (8)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 2 (2)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Social anxiety disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Trichotillomania (Psychiatric disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 9 (10) | 7 (7)
Headache (Nervous system disorders) | 323 (878) | 291 (828)
Idiopathic intracranial hypertension (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 3 (3)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Migraine without aura (Nervous system disorders) | 0 (0) | 1 (1)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 3 (4) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (3) | 3 (3)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2)
Retinal tear (Eye disorders) | 0 (0) | 1 (2)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (6)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (5)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 15 (15)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (6) | 5 (5)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 8 (8) | 4 (4)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (6)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 5 (5)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malpositioned teeth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 132 (260) | 124 (256)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 4 (4) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3)
Ulcerative Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Uvulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (7)
Acne (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 71 (131) | 78 (148)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ligament laxity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 139 (265) | 113 (247)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 2 (3) | 1 (1)
Hypermobility syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Administration site erythema (General disorders) | 53 (139) | 30 (63)
Administration site induration (General disorders) | 54 (136) | 40 (143)
Administration site pain (General disorders) | 524 (2656) | 455 (1949)
Administration site swelling (General disorders) | 49 (136) | 37 (93)
Chest pain (General disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 2 (2) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 318 (974) | 293 (1006)
Influenza like illness (General disorders) | 2 (2) | 6 (6)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 2 (2)
Injection site mass (General disorders) | 0 (0) | 1 (1)
Injection site nodule (General disorders) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 2 (2) | 5 (5)
Injection site pruritus (General disorders) | 1 (1) | 2 (2)
Injection site rash (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 24 (39) | 16 (33)
Swelling face (General disorders) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 2 (2)
Vaccination site reaction (General disorders) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0)
Antinuclear antibody positive (Investigations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 4 (4)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Face injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Immunisation reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (8) | 7 (7)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radial head dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radial nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splinter (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Torus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Underdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Physical assault (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT04707391/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT04707391/SAP_002.pdf